CLINICAL TRIAL: NCT03827655
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Dose Ranging Study to Evaluate the Efficacy and Safety of 2 Dose Regimens of Intravenous TAK-954 for the Prophylaxis and Treatment of Postoperative Gastrointestinal Dysfunction in Patients Undergoing Large- and Small-Bowel Resection
Brief Title: A Study of TAK-954 to Treat Gastrointestinal Dysfunction in Adults After Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-954-2004; 2018-003318-42 (EudraCT Number); U1111-1222-4784 (Registry Identifier: WHO)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Gastrointestinal Dysfunction
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): TAK-954 placebo-matching, 60-minute infusion, intravenously (IV), once presurgery on Day 1 and once daily postsurgery until return of upper and lower GI function or for up to 10 days.
  Interventions: Drug: TAK-954 Placebo
- TAK-954 0.1 mg/100 mL (Experimental): TAK-954 0.1 milligrams per 100 milliliters (mg/100 mL), 60-minute infusion, IV, once presurgery on Day 1 and once daily postsurgery until return of upper and lower GI function or for up to 10 days.
  Interventions: Drug: TAK-954
- TAK-954 0.5 mg/100 mL (Experimental): TAK-954 0.5 mg/100 mL, 60-minute infusion, IV, once presurgery on Day 1 and once daily postsurgery until return of upper and lower GI function or for up to 10 days.
  Interventions: Drug: TAK-954
- TAK-954 0.1 mg/100 mL + Placebo (Experimental): TAK-954 0.1 mg/100 mL, 60-minute infusion, IV, once presurgery on Day 1 and once daily placebo infusions postsurgery up to Day 10 or until resolution of upper and lower GI function.
  Interventions: Drug: TAK-954 Placebo; Drug: TAK-954
- TAK-954 0.5 mg/100 mL + Placebo (Experimental): TAK-954 0.5 mg/100 mL, 60-minute infusion, IV, once presurgery on Day 1 and once daily placebo infusions postsurgery up to Day 10 or until resolution of upper and lower GI function.
  Interventions: Drug: TAK-954 Placebo; Drug: TAK-954

INTERVENTIONS:
Drug: TAK-954 Placebo — TAK-954 placebo-matching intravenous infusion.
  Arms: Placebo; TAK-954 0.1 mg/100 mL + Placebo; TAK-954 0.5 mg/100 mL + Placebo
Drug: TAK-954 — TAK-954 intravenous infusion.
  Arms: TAK-954 0.1 mg/100 mL; TAK-954 0.1 mg/100 mL + Placebo; TAK-954 0.5 mg/100 mL; TAK-954 0.5 mg/100 mL + Placebo

SUMMARY:
The main aim of this study is to check for side effects from TAK-954 and whether it speeds up the recovery of gastrointestinal function after small-bowel or large-bowel resection surgery.

Participants will be treated with TAK-954 before surgery and up to 10 days after surgery.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. In this study TAK-954 is being administered presurgery to evaluate if it can enhance the recovery of GI function postsurgery in participants undergoing open or laparoscopic-assisted partial small- or large-bowel resection. In addition, some participants will also receive TAK-954 postoperatively to evaluate if there is an additional benefit when this drug is administered both pre and post-surgery.

The study will enroll approximately 180 participants. Participants will be equally randomized into one of the three remaining parallel treatment arms- which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

All participants will be given intravenous infusion preoperation and daily postoperation until return of upper and lower GI function or for up to 10 days.

This multi-center trial will be conducted in the United States and Germany. The overall time to participate in this study is up to 100 days. Participants will be treated with the study drug for up to 10 days after surgery or until return of GI function post-surgery (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is scheduled to undergo a laparoscopic-assisted or open partial small- or large-bowel resection.
2. Participant's American Society of Anesthesiologists (ASA) physical status classification is ASA 1 to 3.

Exclusion Criteria:

1. Has significant mechanical bowel obstruction that is not expected to resolve after the surgery, short bowel syndrome, pre-existing clinically significant GI motility disorder (example, gastroparesis, scleroderma, chronic intestinal pseudo-obstruction), uncontrolled diabetes (glycosylated hemoglobin [HbA1c] greater than [>] 10 percent [%]), has an active gastric pacemaker, or requires parenteral nutrition.
2. Had previous major abdominal surgery (example, gastrectomy, gastric bypass, gastric sleeve, lap banding, Whipple, pancreatic resection, total/subtotal colectomy, hemicolectomy, extensive bowel resection).
3. Had a history of radiation therapy to the abdomen or pelvis.
4. Scheduled to undergo any of the following surgeries: low anterior resection, total or subtotal colectomy, colostomy, ileostomy or reversal of stoma, or has a diagnosis that requires rectal resection (eg, tumors in the anorectum) and will likely require lower anterior resection surgery. Participants with planned surgery for which there is no anticipated significant rectal resection and is, therefore, likely to preserve anorectal function and continence postsurgery, will likely be eligible for inclusion in the study if they meet all the study inclusion/exclusion criteria (eg, participants with lesions not involving the rectum [sigmoid colon and above]).
5. Has pre-existing hepatic disease that meets Child-Pugh Class B (moderate; total score 7 to 9 points) or C (severe; total score 10 to 15 points).
6. Has received alvimopan, erythromycin, prucalopride, metoclopramide, domperidone, cisapride, mosapride, renzapride, or azithromycin in the 24 hours prior to starting study drug.
7. Participant has known COVID-19 infection, or suspected COVID-19 infection.
8. Scheduled for abdominal surgery that is classified as emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (25):
- United States (19):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Keck School of Medicine, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Parkview Community Hospital Medical Center, Riverside, California
  - University of Colorado, Aurora, Colorado
  - University of Miami Leonard M. Miller School of Medicine, Miami, Florida
  - Center for Colon & Rectal Surgery - Altamonte Springs, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Stony Brook University Hospital, Stony Brook, New York
  - Fairview Hospital, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - HD Research Corp., Houston, Texas
  - North Star Medical, Houston, Texas
- Germany (6):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Rechts der Isar der Technischen Universitat Munchen, München, Bavaria
  - Universitaetsklinikum Regensburg, Regensburg, Bavaria
  - Sankt Josef-Hospital, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603a4db2bf003ab4a2cf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in Germany and the United States from 07 March 2019 to 27 May 2022.
Pre-assignment Details: Participants with a diagnosis of postoperative gastrointestinal dysfunction were enrolled in a 1:1:1:1:1 ratio into one of the five treatment groups to receive TAK-954 and/or placebo before and after surgery.
Groups:
- Placebo: TAK-954 placebo-matching, 60-minute infusion, intravenously (IV), once presurgery on Day 1 and once daily postsurgery until return of upper and lower gastrointestinal (GI) function or for up to 10 days.
Period: Overall Study
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Started | 52 | 27 | 51 | 27 | 52
Safety Set (Safety Set included all participants who were randomized and received at least 1 dose of double-blind study medication.) | 49 | 26 | 48 | 25 | 50
Full Analysis Set (FAS) (FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid postbaseline on-treatment primary efficacy evaluation (bowel movement or tolerating solid food).) | 45 | 23 | 42 | 21 | 44
Pharmacokinetic (PK) Analysis Set (PK Analysis Set included all participants who were randomized, received at least 1 dose and had at least 1 measurable post-dose plasma for TAK-954.) | 0 | 26 | 47 | 24 | 50
Completed | 45 | 24 | 47 | 25 | 49
Not Completed | 7 | 3 | 4 | 2 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 0 | 1
Not completed — Reason not Specified | 3 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized in the study.
Groups:
- Placebo: TAK-954 placebo-matching, 60-minute infusion, IV, once presurgery on Day 1 and once daily postsurgery until return of upper and lower GI function or for up to 10 days.
- TAK-954 0.1 mg/100 mL: TAK-954 0.1 mg/100 mL, 60-minute infusion, IV, once presurgery on Day 1 and once daily postsurgery until return of upper and lower GI function or for up to 10 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo | Total
Number analyzed (Participants) | 52 | 27 | 51 | 27 | 52 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.99) | 55.9 (13.83) | 57.3 (14.10) | 53.7 (12.15) | 53.2 (15.28) | 55.8 (13.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 10 | 21 | 12 | 26 | 101
  Male | 20 | 17 | 30 | 15 | 26 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 2 | 3 | 10
  Not Hispanic or Latino | 43 | 21 | 37 | 21 | 39 | 161
  Unknown or Not Reported | 8 | 5 | 11 | 4 | 10 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 2 | 0 | 4 | 3 | 14
  White | 37 | 18 | 42 | 18 | 38 | 153
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 9 | 5 | 11 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 8 | 5 | 9 | 4 | 10 | 36
  United States | 44 | 22 | 42 | 23 | 42 | 173
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed is the number of participants with data available for analysis at Baseline.
  centimeters (cm)
    number analyzed (Participants) | 49 | 25 | 47 | 25 | 50 | 196
    (all) | 170.83 (10.991) | 173.01 (9.273) | 172.30 (9.335) | 172.23 (10.972) | 172.60 (9.603) | 172.09 (9.972)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number analyzed is the number of participants with data available for analysis at Baseline.
  kilograms (kg)
    number analyzed (Participants) | 49 | 25 | 47 | 25 | 50 | 196
    (all) | 87.25 (19.317) | 82.92 (18.066) | 87.26 (15.995) | 82.84 (26.018) | 85.64 (20.416) | 85.73 (19.587)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — BMI=[weight(kg)]/[height(m^2)] Population: Number analyzed is the number of participants with data available for analysis at Baseline.
  kilograms per square meter (kg/m^2)
    number analyzed (Participants) | 49 | 25 | 47 | 25 | 50 | 196
    (all) | 29.84 (5.920) | 27.80 (6.492) | 29.45 (5.465) | 27.60 (6.904) | 28.76 (6.652) | 28.93 (6.206)

OUTCOME MEASURES:

1. Primary Outcome: Time From End of the Surgery to Resolution of Upper and Lower Gastrointestinal (GI) Function Postsurgery as Assessed by the Investigator
Description: The time from end of surgery to tolerance of solid food, without first occurrence of vomiting or clinically significant nausea for 1 calendar day after a solid meal (upper GI function) and first spontaneous bowel movement (lower GI function), whichever occurred later up to 10 days postsurgery was observed. Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to Day 10 postsurgery
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid postbaseline on-treatment primary efficacy evaluation (bowel movement or tolerating solid food).
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 1.89 [1.41 to 5.79] | 2.76 [1.51 to 7.85] | 2.59 [0.85 to 4.97] | 2.62 [1.13 to 7.59] | 2.58 [1.46 to 7.74]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.649, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 0.92, 90% CI 2-sided [0.63 to 1.33] — Hazard ratios, 90% confidence intervals (CIs) and associated Wald Chi-square p-values between TAK-954 dose levels and placebo were obtained using a stratified Cox proportional hazard model with treatment as the only independent variable
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.505, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.00, 90% CI 2-sided [0.69 to 1.43] — Hazard ratios, 90% CIs and associated Wald Chi-square p-values between TAK-954 dose levels and placebo are obtained using a stratified Cox proportional hazard model with treatment as the only independent variable

2. Secondary Outcome: Time From the End of the Surgery (Time the Incision is Closed) Until Ready for Discharge as Assessed by the Investigator
Description: The time from the end of surgery (time the incision is closed) until ready for discharge was defined as time from end of surgery until the participant presented effective intestinal transit (spontaneous bowel movement), tolerated solids without vomiting or clinically significant nausea for 1 calendar day after a solid meal, had satisfactory pain control with oral analgesics, and was medically stable/free of complications. Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to Day 24
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 2.03 [1.41 to 16.83] | 2.82 [1.51 to 9.68] | 2.69 [0.85 to 8.79] | 2.94 [1.47 to 7.73] | 2.77 [1.51 to 7.74]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.449, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.03, 90% CI 2-sided [0.71 to 1.49] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.507, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.00, 90% CI 2-sided [0.69 to 1.44] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Time From the End of Surgery Until the Discharge Order is Written
Description: Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to Day 24
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 2.86 [1.62 to 16.72] | 3.95 [1.88 to 10.89] | 2.81 [0.89 to 11.09] | 2.94 [1.47 to 7.81] | 3.33 [1.56 to 14.74]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.406, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.05, 90% CI 2-sided [0.73 to 1.52] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.880, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 0.77, 90% CI 2-sided [0.54 to 1.11] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Time From the End of Surgery to Discharge From Hospital
Description: Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to Day 24
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 2.96 [1.72 to 16.76] | 4.06 [1.97 to 10.89] | 2.89 [1.00 to 11.11] | 3.05 [1.58 to 7.83] | 3.39 [1.70 to 14.77]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.446, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.03, 90% CI 2-sided [0.72 to 1.48] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.892, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 0.76, 90% CI 2-sided [0.53 to 1.09] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Time From End of Surgery to Tolerance of Solid Food as Assessed by the Investigator
Description: The time from end of surgery to tolerance of solid food was defined as intake of solids without vomiting or clinically significant nausea for 1 calendar day after a solid meal. Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to Day 10 postsurgery
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 1.82 [1.41 to 5.79] | 2.76 [1.51 to 7.85] | 2.36 [0.74 to 4.97] | 2.15 [1.13 to 7.59] | 2.55 [1.32 to 7.74]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.760, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 0.86, 90% CI 2-sided [0.60 to 1.23] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.810, Wald chi-squared test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 0.83, 90% CI 2-sided [0.58 to 1.18] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Time From End of Surgery to First Spontaneous Bowel Movement as Assessed by the Investigator
Description: The time from end of surgery to first spontaneous bowel movement was defined as a stool not induced by the use of enemas or laxatives. Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to Day 10 postsurgery
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 1.56 [0.16 to 7.89] | 1.73 [0.11 to 3.81] | 1.11 [0.08 to 4.82] | 1.72 [0.20 to 3.23] | 1.74 [0.53 to 4.94]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.288, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.13, 90% CI 2-sided [0.78 to 1.64] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.453, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.03, 90% CI 2-sided [0.72 to 1.47] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Percentage of Participants With Postoperative Gastrointestinal Dysfunction (POGD) >= 5 Days as Assessed by the Investigator
Description: Participants unable to tolerate solid foods, take anything by mouth, or requiring insertion or reinsertion of nasogastric (NG) tube at or after 5 days post-surgery. Percentages are rounded off to whole number at the nearest single decimal. Stratified Miettinen and Nurminen approach was used for analysis.
Time Frame: Day 1 (surgery) up to Day 10
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
percentage of participants | 8.9 | 8.7 | 2.4 | 4.8 | 9.1
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.046, Stratified Miettinen and Nurminen — P-value was derived using a one-sided test with Ha: Risk Difference<0; Risk Difference (RD) = -0.09, 90% CI 2-sided [-0.17 to 0.00] — The p-values, risk differences and corresponding 90% CIs were obtained using a stratified Miettinen and Nurminen approach with strata weighting by sample size
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.516, Stratified Miettinen and Nurminen — P-value was derived using a one-sided test with Ha: Risk Difference<0; Risk Difference (RD) = 0.00, 90% CI 2-sided [-0.11 to 0.11] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants Requiring Insertion of Nasogastric (NG) Tube Postsurgery
Description: Participants who required insertion of NG tube postsurgery for drainage and symptom relief in case of persistent nausea and vomiting postsurgery were observed. Percentages are rounded off to whole number at the nearest single decimal. Stratified Miettinen and Nurminen approach was used for analysis.
Time Frame: Day 1 (surgery) up to Day 24 postsurgery (10 days of treatment period postsurgery plus 14-day observation period post last dose for recurrence of symptoms)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
percentage of participants | 8.9 | 0.0 | 4.8 | 4.8 | 11.4
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.296, Stratified Miettinen and Nurminen — P-value was derived using a one-sided test with Ha: Risk Difference<0; Risk Difference (RD) = -0.03, 90% CI 2-sided [-0.12 to 0.06] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.677, Stratified Miettinen and Nurminen — P-value was derived using a one-sided test with Ha: Risk Difference<0; Risk Difference (RD) = 0.03, 90% CI 2-sided [-0.07 to 0.13] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Time From End of Surgery to First Flatus
Description: Kaplan-Meier survival analysis method was used.
Time Frame: Day 1 (surgery) up to first flatus (up to Day 10 postsurgery)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Groups:
- Placebo: TAK-954 placebo-matching, 60-minute IV, once presurgery on Day 1 and once daily postsurgery until return of upper and lower GI function or for up to 10 days.
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 45 | 23 | 42 | 21 | 44
days | 1.21 [0.06 to 6.22] | 1.26 [0.28 to 7.62] | 0.96 [0.08 to 3.04] | 1.18 [0.20 to 2.82] | 1.12 [0.02 to 3.88]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.5 mg/100 mL; Test type: Superiority; p = 0.338, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.10, 90% CI 2-sided [0.76 to 1.57] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.5 mg/100 mL + Placebo; Test type: Superiority; p = 0.422, Wald chi-square test — P-values were derived using a one-sided test with alternative hypothesis (Ha): Hazard Ratio>1; Hazard Ratio (HR) = 1.04, 90% CI 2-sided [0.73 to 1.49] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Observed Plasma Concentration of TAK-954 at the End of Infusion on Day 1
Time Frame: Day 1 (surgery): postinfusion
Population: PK Analysis Set included all participants who were randomized, received at least 1 dose and had at least 1 measurable post-dose plasma for TAK-954. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
Number analyzed (Participants) | 20 | 33 | 20 | 35
picograms per milliliter (pg/mL) | 1190 (480) | 5220 (1810) | 2500 (4140) | 12000 (28500)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 100
Description: All-cause Mortality: All participants enrolled in the study. Serious and Other Adverse Events: Safety Set included all participants who were randomized and received at least 1 dose of double-blind study medication.
Arm/Group | Placebo | TAK-954 0.1 mg/100 mL | TAK-954 0.5 mg/100 mL | TAK-954 0.1 mg/100 mL + Placebo | TAK-954 0.5 mg/100 mL + Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/27 | 0/51 | 0/27 | 1/52
Serious Adverse Events (participants affected / at risk) | 8/49 | 9/26 | 8/48 | 2/25 | 11/50
Other Adverse Events (participants affected / at risk) | 46/49 | 23/26 | 39/48 | 21/25 | 41/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | TAK-954 0.1 mg/100 mL (N=26) | TAK-954 0.5 mg/100 mL (N=48) | TAK-954 0.1 mg/100 mL + Placebo (N=25) | TAK-954 0.5 mg/100 mL + Placebo (N=50)
Abdominal abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dehiscence (General disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 5
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Urinoma (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | TAK-954 0.1 mg/100 mL (N=26) | TAK-954 0.5 mg/100 mL (N=48) | TAK-954 0.1 mg/100 mL + Placebo (N=25) | TAK-954 0.5 mg/100 mL + Placebo (N=50)
Abdominal distension (Gastrointestinal disorders) | 5 | 1 | 5 | 1 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 7 | 1 | 6 | 2 | 4
Anaemia postoperative (Injury, poisoning and procedural complications) | 6 | 1 | 9 | 2 | 5
Bradycardia (Cardiac disorders) | 3 | 0 | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 11 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 2 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 1 | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 0 | 3
Hypertension (Vascular disorders) | 6 | 1 | 7 | 0 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 1 | 10 | 1 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5 | 2 | 4 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 4 | 3 | 1 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5 | 3 | 1 | 4
Hypotension (Vascular disorders) | 3 | 0 | 4 | 0 | 4
Leukocytosis (Blood and lymphatic system disorders) | 6 | 1 | 4 | 0 | 4
Nausea (Gastrointestinal disorders) | 22 | 14 | 20 | 12 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 3
Postoperative ileus (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 5 | 0 | 4 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 15 | 0 | 9 | 0 | 10
Procedural nausea (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 4 | 5 | 2 | 4 | 4
Pyrexia (General disorders) | 3 | 3 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 1 | 2 | 0 | 3
Urinary retention (Renal and urinary disorders) | 4 | 3 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Urine output decreased (Investigations) | 1 | 0 | 2 | 0 | 3
Vomiting (Gastrointestinal disorders) | 14 | 8 | 8 | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03827655/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03827655/SAP_001.pdf